CLINICAL TRIAL: NCT06029985
Title: Long-term Follow up of the Cases Who Underwent Conservative Surgery for Placenta Previa Accreta: a Prospective Case Series Study
Brief Title: Hysteroscopic Follow-up Following Conservative Stepwise Surgical Approach for Management of Placenta Previa Accreta
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Mahmoud Mohamed Ghaleb, Professor, Ain Shams Maternity Hospital
Other Study IDs: Hysteroscopic Follow-Up
Record Dates: First submitted 2023-08-26; First posted 2023-09-08 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hysteroscopic Follow Up — Office hysteroscopy was carried out to detect the scar site, performed with a 4-mm, continuous-flow operative hysteroscope by vaginoscopic approach, without analgesia or anesthesia. Distension of the uterus was obtained using a normal solution as distension medium, dispensed by an electronic suction/irrigation pump. This can maintain a constant intrauterine pressure of around 30-40 mmHg, balancing an irrigation flow of 200 mL/min with a vacuum of 0.2 bars, necessary to avoid overdistension of the muscle fibers and patient discomfort. The use of this distension medium allows blood or mucus to be washed out from the pouch if necessary.

SUMMARY:
Conservative management of placenta accreta spectrum can preserve future fertility but should only be done in hospitals with enough experience as it carries a high risk of maternal complications.

Follow up after conservative management is crucial to detect complications early.

DETAILED DESCRIPTION:
Placenta accreta is defined histopathologically as abnormal trophoblast invasion of part or all of the placenta into the myometrium of the uterine wall.1 Depending on the depth of villous tissue invasiveness, placenta accreta was subdivided by pathologists into "creta", "increta", and "percreta", in which the villi adhere superficially to the myometrium without interposing decidua, penetrate deeply into the uterine myometrium, and perforate through the entire uterine wall and may invade the surrounding pelvic organs, respectively.

The term placenta accreta spectrum (PAS) will be used in this manuscript to include both the abnormally adherent and the invasive forms of accreta placentation. Severe and sometimes life-threatening hemorrhage, which often requires blood transfusion, increases maternal morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women with one or more previous cesarean deliveries
2. Women diagnosed with placenta previa accreta and underwent Conservative stepwise surgical approach for management.

Exclusion Criteria:

1. women who refused to participate in the study.
2. Associated other medical conditions as pregnancy-induced hypertension, heart diseases, and rheumatological diseases apart from iron deficiency anemia.
3. Presence of uterine anomalies

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Women with one or more previous cesarean deliveries who were diagnosed with placenta previa accreta and underwent Conservative stepwise surgical approach for management in Ain shams maternity hospital
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Easiness of hysteroscopy introduction | 3-6 months
  accessibility of hysteroscopic examination
Adequacy of uterine cavity | 3-6 months
  visualization of the uterus will be assessed using office hysteroscopy
intrauterine adhesions | 3-6 months
  visualization of the intrauterine adhesions will be assessed using office hysteroscopy
cesarean scar niche | 3-6 months
  presence of a pouch, that forms on the wall of your uterus.
Menstrual pattern | 3-6 months
  menstrual irregularities by history regarding Regular and normal volume or Regular and scanty or presence of Intermenstrual bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Samy, MD, Study Director — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No